CLINICAL TRIAL: NCT04064190
Title: A Phase 2 Study of TGF-β Inhibition (Vactosertib) with Anti-PD-L1 (Durvalumab) in Patients with Advanced or Recurrent Urothelial Carcinoma Failing to Achieve Response with Checkpoint Inhibition
Brief Title: Vactosertib with Durvalumab in Urothelial Carcinoma Failing Checkpoint Inhibition
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changing trial strategy
Sponsor: MedPacto, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-VAC-202
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Urothelial Carcinoma Recurrent; Advanced Urothelial Carcinoma
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Phase 2, open label, non randomized single arm study with two cohorts and a safety run-in for first six patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vactosertib+Durvalumab (Experimental): Vactosertib will be administered in combination with standard dose of durvalumab every four weeks.
  Interventions: Drug: Vactosertib(TEW-7197)/ Durvalumab

INTERVENTIONS:
Drug: Vactosertib(TEW-7197)/ Durvalumab — Vactosertib (PO) in combination with Durvalumab (IV) every 4 weeks

SUMMARY:
This is Phase 2, open label, non randomized single arm study to determine whether the administration of vactosertib with durvalumab will provide meaningful increases in the Overall Response Rate (ORR) in patients with urothelial cancers that fail to achieve a response with anti-PD-1/PD-L1 based regimens

DETAILED DESCRIPTION:
This is a Phase 2, open-label, non-randomized, two-cohort multi center study with a safety run-in of 6 patients in Cohort 1. It is anticipated that a total of 48 patients will be enrolled.

Durvalumab will be administered with the standard regimen of 1500 mg intravenously (IV) every four weeks. Vactosertib will be administered at a dose of 300 mg PO BID for 5 days per week All treatment will be administered up to two years and the trial is anticipated to be completed over a period of 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at enrollment
2. Histologically or cytologically documented locally advanced/inoperable or metastatic urothelial bladder carcinoma (UBC), including renal pelvis, ureters, urinary bladder, and urethra.
3. Prior anti-PD-(L)1 treatment.
4. Measurable disease per RECIST 1.1 assessed by computed tomography (CT) scan or MRI.
5. Recurrent disease after any prior platinum-based chemotherapy regimen or ineligible for platinum therapy.
6. Adequate organ and marrow function as defined
7. Must have a life expectancy of at least 12 weeks.
8. Body weight > 30 kg

Exclusion Criteria:

1. History of allogeneic organ transplantation.
2. Active or prior documented autoimmune or inflammatory disorders
3. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure .
4. History of another primary malignancy
5. History of leptomeningeal carcinomatosis.
6. History of active primary immunodeficiency.
7. Active infection including tuberculosis, hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus .
8. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 12months
  ORR by RECIST version 1.1

SECONDARY OUTCOMES:
Time to Tumor Response | Overall study period up to 3years
  TTR by RECIST version 1.1 and iRECIST
Best Response | Overall study period up to 3years
  Best response (percent of tumor shrinkage) by RECIST version 1.1 and iRECIST
Duration of Response | Overall study period up to 3years
  DoR by RECIST version 1.1 and iRECIST
Progression Free Survival | 6-month/ 12-month
  PFS by RECIST version 1.1 and iRECIST
Overall survival | 12month
  OS by RECIST version 1.1 and iRECIST
Tumor-specific immune responses | Overall study period up to 3years
  tumor-specific immune responses within on-therapy biopsies measured by increased T cell infiltration and increased IFN-λ signature. and the correlation with outcome as measured by ORR, TTR, DoR, PFS and OS
Incidence of Treatment-Emergent Adverse Events [Safety and tolerability] | Overall study period up to 3years
  To assess safety and tolerability of vactosertib administered concurrent with Durvalumab in patients with urothelial carcinoma failing checkpoint inhibition

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No